CLINICAL TRIAL: NCT07384052
Title: Safety and Feasibility of Intranasal Insulin in Patients With Spinal Cord Injury
Acronym: INI-SCI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Department of Defense Congressionally Directed Medical Research Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: A22-210-01; CDMRP-SC220220 (Other: Department of Defense Congressionally Directed Medical Research Program)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury
Keywords: Insulin; Intranasal; Safety; Feasibility; Spinal Cord Injury; SCI; INI
MeSH Terms: conditions — Spinal Cord Injuries; Insulin Resistance | interventions — Insulin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of 2 groups: 76 IU insulin, or saline (placebo) control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Insulin (Experimental): Regular Insulin (Novolin-R) 76 international units per day administered as 38 IU in one nostril twice daily (alternating nostrils) for 21+/-3 days
  Interventions: Drug: Regular Insulin
- Placebo (Placebo Comparator): 0.9% sodium chloride in one nostril twice daily (alternating nostrils) for 21+/- days
  Interventions: Other: 0.9 % Normal Saline

INTERVENTIONS:
Drug: Regular Insulin — Administered Intranasally at 76 IU
  Other Names: Novolin-R
  Arms: Intranasal Insulin
Other: 0.9 % Normal Saline — Placebo Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether insulin, a drug approved by the FDA for the treatment of diabetes mellitus, is safe when administered as a nasal spray (intranasally) to people who have experienced a spinal cord injury. While insulin nasal spray has been shown to be safe in many patient populations, it has not yet been studied in people with spinal cord injury. This study would be the first step to developing insulin nasal spray as a treatment for spinal cord injury in the future.

This study is recruiting up to 12 individuals who have experienced a spinal cord injury at least 4 months ago to administer either 76 IU insulin nasal spray or a placebo (inactive nasal spray) at home every day for up to 24 days. Participants will be asked questions about their health and symptoms related their spinal cord injury, and will have their blood collected throughout the study. Participants who are unable to administer the medication independently must have a study partner in order to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 and <85 years of age
2. Subject has sustained a traumatic or non-traumatic spinal cord injury with American Spinal Injury Association (ASIA) rating A, B, C or D, complete or incomplete
3. Subject sustained spinal cord injury at least 4 months before baseline visit
4. Female subjects must have either: (1) a negative pregnancy test at the screening and treatment visits OR (2) be at least 2 years post-menopausal / surgically sterile
5. The subject must be proficient in English in order to comply with instructions and measures for the study
6. Subject is able to prepare and administer the study drug as outlined in the protocol or has a carer who is available to do so for the duration of the study
7. Subject can provide written informed consent
8. Subject has been on a stable regimen of medications for at least 30 days from baseline visit

Exclusion Criteria:

1. Subject is dependent on a ventilator or has a patent tracheostomy site
2. Subject has recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a sudden rise in systolic BP greater than 20 mmHg or diastolic BP greater than 10 mmHg without rise in heart rate and accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, or blurry vision
3. Subject has medical history and/or clinically determined disorders: chronic sinusitis, previous nasal and/or oto-pharyngeal surgery and severe deviated septum and/or other anomalies
4. Subject has history of any of the following: active and significant central nervous system, psychiatric illness, pulmonary, or cardiovascular disorders or any other clinically relevant abnormality that inclusion would pose a safety risk to the subject as determined by investigator
5. Subject has participated in a clinical trial investigation within 3 months of this study
6. Subject has a history of allergy, hypersensitivity, or other significant adverse reaction to insulin
7. Subject is taking insulin for Type I or Type II diabetes
8. Subject is pregnant or breast feeding
9. Any other clinically relevant finding that would pose a safety risk to the subject as determined by the investigator

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety measured by number of serious adverse events (SAE) and adverse events (AE) | 3 weeks
  Total number of AEs/SAEs during the course of treatment. More AEs/SAEs indicates a less safe treatment. AEs counts will include total count and will be stratified by severity.

SECONDARY OUTCOMES:
Treatment adherence as assessed by participant Daily Drug Diaries | 3 weeks
  Number of doses successfully administered as reported by participants in their daily drug diaries
Feasibility of virtual training as assessed by the Virtual Training Compliance Checklist | Baseline Visit
  Average score on virtual training compliance checklist, both arms combined
Acceptability of virtual training as assessed by the Virtual Training and Feasibility and Acceptability Survey | Baseline
  Total score on the Virtual Training Feasibility and Acceptability Survey, both arms combined
Feasibility of blood spot collection procedure as measured by a Blood Spot Procedure Compliance Checklist | Screening Visit
  Participants will be trained to perform a blood spot collection procedure independently. Feasibility will be measured by the average score on blood spot procedure compliance checklist, both arms combined
Acceptability of Blood Spot Procedure, as measured by a Blood Spot Procedure Post-Training Acceptability Survey | Screening Visit
  Acceptability of performing blood spot procedure independently will be measured by the average score on a blood spot procedure post-training acceptability survey, both arms combined

CONTACTS AND LOCATIONS:
Overall Officials: Leah R Hanson, PhD, Principal Investigator — HealthPartners Institute; Kimberly Byrnes, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided